CLINICAL TRIAL: NCT03255538
Title: Deep Friction Massage Effects on Pain and Function in Patellar Tendinopathy
Brief Title: Deep Friction Massage: Symptomatic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Responsible Party: Principal Investigator, Maria Paço, PhD, Clinical research, Cooperativa de Ensino Superior, Politécnico e Universitário
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DFM_2
Record Dates: First submitted 2017-08-18; First posted 2017-08-21 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Tendinopathy
Keywords: patellar tendon
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DFM: Mean pressure (Experimental): In this group, deep friction massage will be applied with the mean pressure, previously obtained in a baseline assessment.
  Interventions: Other: DFM: Mean pressure
- DFM: Mean pressure - 25% (Experimental): In this group, deep friction massage will be applied will less 25% of the pressure previously obtained in a baseline assessment.
  Interventions: Other: DFM: Mean pressure - 25%
- DFM: Mean pressure +25% (Experimental): In this group, deep friction massage will be applied will an increment of 25% of the pressure previously obtained in a baseline assessment.
  Interventions: Other: DFM: Mean pressure + 25%
- Control session (No Intervention): In this group, the participants will rest for 15 minutes

INTERVENTIONS:
Other: DFM: Mean pressure — Deep friction massage as described by Dr. James Cyriax, performed with the mean pressure previously obtained in a baseline assessment.
  Arms: DFM: Mean pressure
Other: DFM: Mean pressure - 25% — Deep friction massage as described by Dr. James Cyriax, performed with the mean pressure previously obtained in a baseline assessment decremented by 25%.
  Arms: DFM: Mean pressure - 25%
Other: DFM: Mean pressure + 25% — Deep friction massage as described by Dr. James Cyriax, performed with the mean pressure previously obtained in a baseline assessment incremented by 25%.
  Arms: DFM: Mean pressure +25%

SUMMARY:
Despite DFM being a widely-used technique and the empirical grounding regarding the importance of the pressure applied, there is no study characterizing the pressure applied during DFM, remaining it a discretion of the physiotherapist. Additionally, it is not known how the amount of pressure applied may influence pain mechanisms or function in the symptomatic patellar tendon. Having this, our objective is to characterize the pressure applied during deep friction massage and evaluate the immediate effects of different pressures applied during deep friction massage in the time until analgesia as well as in function, in patellar tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* The participants should have a symptomatic patellar tendon

Exclusion Criteria:

* History of other previous injuries of the lower limbs;
* Intake of medication that could interfere with pain mechanisms;
* Presence of any factors or conditions that could interfere with the awareness and sensibility to pain.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Time until analgesia | 10 minutes
  Time until self reported sensation of analgesia, controlled by a chronometer, since the application of deep friction massage.
Numeric Pain Rating Scale | 20 minutes
  Self-reported pain intensity.
Maximal isometric strength of quadriceps | 20 minutes
  Measure of maximal isometric strength, through a dynamometer.
Knee flexion range of movement | 20 minutes
  Measure of knee flexion range of movement, through a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Paço, PhD, Principal Investigator — Cooperativa Ensino Superior Politécnico e Universitário
Locations (1):
- Cooperativa Ensino Superior Politécnico e Universitário, Gandra, Paredes, Portugal

IPD SHARING:
Plan to Share IPD: No